NCT05933252

MDAnderson Cancer Center Study Number: 2023-0097

May 07, 2024 Page 1 of 12

## Informed Consent/Authorization for Participation in Research

administering an electronic tool to assess

postoperative pAin, nausea, and Vomiting in English

or Spanish-Speaking pediatric patients with neoplastic conditions: The AVESS Study

**Protocol No.:** 2023-0097

**Sponsor:** National Institute of Drug Abuse

**Investigator:** Juan Cata, MD

STUDY-RELATED

**PHONE NUMBER(s):** 713-582-6452

| Participant's Name | Medical Record Number |
|--------------------|-----------------------|

## **Key Information**

The following is a short summary of this study to help you decide whether or not to be a part of this study. More detailed information is listed later on in this form.

If you are reading and signing this form on behalf of a potential participant, please note: Any time the words "you," "your," "I," or "me" appear, it is meant to apply to the potential participant.

## Why am I being invited to take part in a research study?

You are invited to take part in a research study because you may experience pain after cancer surgery, and doctors would like to study your pain using an augmented reality (AR) application.

# What should I know about a research study?

Someone will explain this research study to you.



- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

### Why is this research being done?

The goal of this pilot research study is to look at the feasibility of using an electronic tool to measure pain, nausea, and vomiting after surgery in English or Spanish-speaking pediatric cancer patients. Augmented reality (AR) lets you view the real world through a device's camera and application ("app") but adds virtual or digital characters and items to the image.

## How long will the research last and what will I need to do?

You are expected to be in this research study until you are discharged from the hospital after surgery.

You will be asked to tell the study team about your pain, nausea, and/or vomiting using an app on an iPad every 15 minutes during your recovery period in the Post-Anesthesia Care Unit (PACU). During the time you are on study, information about your health, pain levels, and use of pain medications will also be collected from your medical record.

More detailed information about the study procedures can be found under "What happens if I agree to be in this research?"

## Is there any way being in this study could be bad for me?

Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment.

More detailed information about the risks of this study can be found under "Is there any way being in this study could be bad for me? (Detailed Risks)"

## Will being in this study help me in any way?

It cannot be promised that there will be any benefits to you or others from your taking part in this research. However, possible benefits include providing a more accurate report of your symptoms, which may help the medical staff treat them better. Future patients may benefit from what is learned. There may be no benefits for you in this study.



## What happens if I do not want to be in this research?

Participation in research is completely voluntary. You can decide to participate, not participate, or discontinue participation at any time without penalty or loss of your regular benefits.

Instead of taking part in this study, you may choose to have standard-of-care surgery without using the AR application in the iPad. This option has risks and benefits that may be the same or different than those in this research study. The study doctor can discuss this option, including its risks and benefits, with you.

## **Detailed Information**

The following is more detailed information about this study in addition to the information listed above.

### Who can I talk to if I have questions or concerns?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team at 713-582-6452.

This research has been reviewed and approved by an Institutional Review Board ("IRB" - an ethics committee that reviews research studies). You may talk to them at (713) 792-6477 or <a href="mailto:IRB">IRB</a> Help@mdanderson.org if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

## How many people will be in this study?

It is expected about 16 people at MD Anderson will be enrolled in this research study.

## What happens if I agree to be in this research?

#### **Post-Surgery Period**

If you agree to take part in this study, you will be given a hospital-issued iPad and asked to use the AR app to measure and record the level of your pain, nausea, vomiting, or retching. The study team will show you how to use the AR app.



You will be asked to report your symptoms every 15 minutes while you are in recovery. You will return the iPad to the study team when you are ready to go to your hospital room.

Every day that you are in the hospital after surgery, the study team will check your medical record to track if you are prescribed opioids/pain medication and how many times you use the pain medication given to you after surgery. You and/or your parent/guardian will be asked how much pain you are feeling as well.

You will not have access to the iPad after you leave the hospital.

#### Data Collection

Information will also be collected from your medical record during the study. This may include demographic information (age, sex, race, date of birth, and so on) and information about your medical history (for example, underlying medical conditions, date of surgery, pain levels, or use of pain medications or other drugs you are taking).

#### **Discharge Questionnaires**

On the day that you leave the hospital (are discharged), you will complete questionnaires about your overall experience with the app and your quality of life. Depending on your age, your guardian/caregiver may complete the questionnaire for you. These questionnaires will take about 10 minutes to complete. Your participation in the study will finish that day.

## What happens if I say yes, but I change my mind later?

You can leave the research at any time; it will not be held against you.

If you decide you want to stop taking part in the study, it is recommended that you first talk to your doctor. If you withdraw from this study, you can still choose to be treated at MD Anderson.

If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can collect data from your routine medical care. If you agree, this data will be handled the same as research data.

# Is there any way being in this study could be bad for me? (Detailed Risks)

You should discuss the risks of **questionnaires** with the study chair. The known risks are listed in this form, but they will vary from person to person. Some questions may make you feel upset or uncomfortable. You may refuse to answer any question. If you have concerns after completing the questionnaire(s), you are encouraged to contact your doctor or the study chair. If you experience significant distress caused by any of the questions in the questionnaire, the study chair, child-life specialist, and/or a psychologist will discuss your concerns with you, if needed.



While you **interact with app in the iPad**, there is a rare (less than 1% chance) risk of falls, dizziness, and/or nausea.

In addition to these risks, this research may hurt you in ways that are unknown. These may be a minor inconvenience or may be more serious.

You will be told about any new information that may affect your health, welfare, or choice to stay in the research.

# Will it cost anything to be in this study? Will I be paid to be in this study?

There is no cost to you for taking part in this study. You and/or your insurance provider will be responsible for the cost of standard-of-care surgery and opioid medications you receive as part of your routine care.

If the iPad is lost or broken during the study, you should report it to the study team. You will not be responsible for the cost of the lost or broken iPad.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

You will not receive any compensation for taking part in this study.

## What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study and medical records, to people who need to review this information. Complete secrecy cannot be promised. Organizations that may inspect and copy your information include the IRB and other representatives of this organization.

Any personal information that could identify you will be removed or changed before data are shared with other researchers or results are made public.

Study data will be collected and managed using REDCap (Research Electronic Data Capture) electronic data capture tools hosted at MD Anderson. REDCap is a secure,



web-based application with controlled access designed to support data capture for research studies.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate DOES NOT stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

The sponsor, monitors, auditors, the IRB, and the Food and Drug Administration will be granted direct access to your medical records to conduct and oversee the research. By signing this document, you are authorizing this access. The results of this research may be published. However, your name and other identifying information will be kept confidential.

Federal law provides additional protections of your medical records and related health information. These are described below.

## Will my data be used for future research?

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson, National Institute of Drug Abuse, or shared with other researchers and/or institutions for use in future research.

In some cases, all of your identifying information may not be removed before your data are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the MD Anderson IRB before your data can be used. At that time, the IRB will decide whether or not further permission from you is required. If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data.



If identifiers are removed from your identifiable private information that is collected during this research, that information could be used for future research studies or shared with another researcher for future research studies without your additional informed consent.

### Can I be removed from the research study without my permission?

The person in charge of the research study or the sponsor can remove you from the research study without your approval. If you are removed from the study early, the study staff will tell you why.

### What happens if I get hurt from being in this study?

If you get sick or hurt and it is related to your participation in this study, you will be given care at MD Anderson (if you are at the clinic when you are sick or hurt). If you get hurt or sick and you are not at the clinic (for example, you are at home or at another doctor's office):

- call your personal doctor right away (or in an emergency, call 911)
- tell your personal doctor or ER staff that you are in this study (try to give them a copy of this consent form or show them your participant card)

If you suffer a study-related injury, you may contact the Chair of the study, Dr. Juan Cata, at 713-582-6452 or 713-792-2121 (24 hours) with any questions you may have.

You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. Costs of treatment received because you were hurt or sick will be billed to you or your insurance company. No other form of payment is available.

You may also call the MD Anderson IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

#### What else do I need to know?

This research is being funded by the National Institute of Drug Abuse.

MD Anderson may benefit from your participation and/or what is learned in this study.

Your information (both identifiable and de-identified) may be used to create products or to deliver services, including some that may be sold and/or make money for others. If this happens, there are no plans to tell you, or to pay you, or to give any compensation to you or your family.



# Authorization for Use and Disclosure of Protected Health Information (PHI):

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - The National Institute of Drug Abuse, who is a sponsor or supporter of this study, and/or any future sponsors/supporters of the study, and/or licensees of the study technology
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants and it may be re-disclosed.

Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.

- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify



MDAnderson

Cancer Center

you. At most, the Web site will include a summary of the results. You can search this Web site at any time.



# CONSENT/AUTHORIZATION (Adult Participants Only)

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document.

| any of my legal rights. I will be given a signed copy of this cons | sent document. |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| PRINTED NAME OF PARTICIPANT | |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or representative, using language that is understandable and appr have fully informed this participant of the nature of this study an and risks and that the participant understood this explanation. | opriate. I believe that |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |



| I have read and understand the description of this research. I have h discuss the study and ask questions. My questions have been answ permission for my child or ward to take part in this study. | |
|---|---|
| SIGNATURE OF PARENT/GUARDIAN | DATE |
| PRINTED NAME OF PARENT/GUARDIAN | |
| SIGNATURE OF PARENT/GUARDIAN Signature of Other Parent (Optional, unless required by the IRB.) | DATE |
| PRINTED NAME OF PARENT/GUARDIAN | |
| The IRB has determined that the signature of both parents is re- | quired. |
| If not obtaining both parental signatures, please indicate reason belo | w: |
| Other parent is deceased, unknown, incompetent, or not reason | ably available. |
| Parent/Guardian signing above has sole legal responsibility for to custody of the child. | the care and |
| X The IRB has determined that the signature of both parents is | NOT required. |
| ASSENT OF MINOR (Entire section must be completed if the participant's intellectual age is at least 18 years. Participants with an intellectual age of 7 - 12 are not required to significant. | |
| If written assent is not obtained on an age-appropriate participant, ch | neck reason why not: |
| 1.) The participant's intellectual age is less than seven. | |
| 2.) The participant dissented, but the participant's parent(s)/gua<br>intervention(s) or procedure(s) involved in the research hold<br>of a direct benefit that is important to the health and/or well<br>participant and is available only in the context of this resear | d out the possibility being of the |
| 3.) Other: | |
| I have been told what I will be asked to do in this study. | |



Cancer Center
I have been told that I do not have to be in this study. If I decide not to be in this study, no one will be mad at me. I may quit at any time, but if I do, I may need to take a different treatment.

| I have had a chance to talk about the study and ask the study doctor<br>my questions have been answered. I agree to be in this study and<br>to do so long as I want to stay in this study. I agree that the study on<br>this study. By signing this paper, I am not giving up any of my le<br>been given a copy of this document. | do what I am asked<br>loctor can put me |
|---|---|
| SIGNATURE OF MINOR (Age 13-17) | DATE |
| DDINTED NAME OF MINOR | |